CLINICAL TRIAL: NCT05225311
Title: Fetal Ebstein Anomaly and Tricuspid Valve Dysplasia Registry
Acronym: FEAT Registry
Status: Recruiting | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Lindsay Freud, Head of Fetal Cardiology, The Hospital for Sick Children
Other Study IDs: 1000076991
Record Dates: First submitted 2022-01-06; First posted 2022-02-04 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Ebstein Anomaly; Tricuspid Valve Dysplasia
MeSH Terms: conditions — Ebstein Anomaly | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Fetal Ebstein's Anomaly or Tricuspid Valve Dysplasia: Patients will be followed for life-long outcomes.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Patients will be followed by the registry for life-long outcomes.

SUMMARY:
Ebstein anomaly and tricuspid valve dysplasia (EA/TVD) are rare congenital tricuspid valve malformations that carry among the highest mortality of all congenital heart disease diagnosed in utero. Despite the high mortality associated with severe EA/TVD in the fetus, it has only been studied retrospectively. By prospectively enrolling a cohort across multiple centers, many questions may be answered in the perinatal period and beyond. The registry will allow us to understand perinatal and postnatal decision-making in this complex group of patients across centers.

Given the rarity of the disease, a retrospective arm was added to the original prospective study in May 2024.

ELIGIBILITY:
Inclusion Criteria:

1. Mothers of fetuses (ages 14-54) diagnosed with EA/TVD of any severity with normal segmental anatomy (AV and VA concordance)

   1. Mothers may be enrolled at any gestational age, up to the day of pregnancy outcome (elective termination of pregnancy, demise, or live-birth)
   2. Singletons, twins or higher order multiples may be included
2. Consent obtained at a participating site

Exclusion Criteria:

1. Mothers of fetuses diagnosed with EA/TVD in the context of abnormal segmental anatomy (AV and/or VA discordance) or other lesions, such as congenitally corrected transposition of the great arteries or pulmonary atresia with intact ventricular septum
2. Unable or unwilling to provide consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Fetuses diagnosed with EA/TVD of any severity with normal segmental anatomy (AV and VA concordance)
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-09-22 (Actual); Primary Completion 2050-09 (Estimated); Study Completion 2055-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of fetuses who survive to live-birth at term | 37 0/7 to 40 0/7 weeks gestation
Proportion of live-born children who survive to 30 days | 0-30 days
Freedom from death beyond the neonatal period | 30 days-30 years

SECONDARY OUTCOMES:
Change in umbilical artery pulsatility index throughout gestation | 20 0/7 to 40 0/7 weeks gestation
Proportion with hydrops throughout gestation | 20 0/7 to 40 0/7 weeks
Average gestational age at birth | At birth
Average birth weight | At birth
Proportion who undergo neonatal cardiac surgery | 0-30 days
Freedom from cardiac re-intervention | 30 days-30 years
Freedom from cardiac arrhythmia | 30 days-30 years
Infant neurodevelopment as assessed by Bayley Scales of Infant Development | 12-15 months
Pediatric neurodevelopment as assessed by Adaptive Behavior Assessment System | 3-18 years
Quality of life as assessed by Peds QL General and Cardiac Modules | 2-30 years

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No